CLINICAL TRIAL: NCT05133050
Title: Safety and Efficacy of Early Angiotensin-converting Enzyme Inhibition in Patients With Alport Syndrome Carrying Pathogenic Heterozygous COL4A3,COL4A4 or COL4A5 Mutations
Brief Title: Safety and Efficacy of ACEI in Alport Syndrome Patients With COL4A3/COL4A4/COL4A5 Variants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2021-070-2
Record Dates: First submitted 2021-10-27; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Alport Syndrome
MeSH Terms: conditions — Nephritis, Hereditary | interventions — Ramipril

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Drug: Ramipril The initial dose of ramipril is 2.5 mg /d. The blood pressure, blood potassium and blood creatinine is measured every 1-2 weeks. If the blood pressure is normal, the dose of ramipril is adjusted to 5 mg /d after 2 weeks. If the blood pressure is low, the dose of ramipril is reduced to 1.25 mg /d until the blood pressure becomes normal, otherwise, stop ramipril using. If the blood potassium is high (>5.5mmol/L), the dose of ramipril is reduced to 1.25 mg /d until the blood potassium becomes normal, otherwise, stop ramipril using. If the blood creatinine is higher before therapy (≥30%), the dose of ramipril is reduced to 1.25 mg /d until the blood creatinine becomes normal, otherwise, stop ramipril using.
  Interventions: Drug: Ramipril
- Control group (No Intervention): No angiotensin converting enzyme inhibitor (ACEI) and other renin-angiotensin system inhibitors (including angiotensin II receptor antagonists, etc.) treatment.

INTERVENTIONS:
Drug: Ramipril — We use ACEI: ramipril, in this prospective, randomized, controlled and multicenter clinical trial to access the safety and efficacy in Alport syndrome patients carried COL4A3/COL4A4/COL4A5 variants.
  Arms: Experimental group

SUMMARY:
Alport syndrome (AS) is the second most common monogenic cause of end-stage renal failure (ESRF). AS is caused by variants in the COL4A3, COL4A4, and COL4A5 genes, which encode for the a3, a4, and a5 chains of type IV collagen. This trial is a prospective, randomized, controlled and multicenter trial. Mainly to assess the safety and efficacy of ramipril in Alport syndrome patients with variants of COL4A3/COL4A4/COL4A5.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30-50 Years;
2. Sex: All;
3. Alport syndrome patients with variants of COL4A3/COL4A4/COL4A5; hematuria or microalbuminuria; eGFR>90 mL/min/1.73m2;
4. Patients with microscopic hematuria only;
5. Patients with microscopic hematuria and microalbuminuria: 30-300mg/24h or urine albumin/creatinine: 30-300mg/g;
6. No angiotensin converting enzyme inhibitor (ACEI) and other renin-angiotensin system inhibitors (including angiotensin II receptor antagonists, etc.) treatment.

Exclusion Criteria:

1. With primary or secondary kidney disease, including IgA nephropathy, membranous nephropathy, lupus nephropathy, benign renal arterioles, etc.;
2. Patients with a history of angioedema;
3. Hypovolemia or hypotension (systolic blood pressure less than 90mmHg and/or diastolic blood pressure less than 60mmHg);
4. Pregnant and lactating women;
5. Patients with bilateral renal artery stenosis or unilateral renal artery stenosis with solitary kidney;
6. Hyperkalemia, blood potassium>5.5mmol/L;
7. Severe aortic stenosis, severe mitral stenosis;
8. Treatment of drug allergy;
9. Hypertension or other diseases that may require treatment with angiotensin-converting enzyme inhibitors;
10. Disagree to participate in this research.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 510 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease progression time | Up to 240 weeks
  a) Patients from no proteinuria to microalbuminuria; b) patients from microalbuminuria to dominant proteinuria.

SECONDARY OUTCOMES:
5-year disease progression rate and eGFR slope | Up to 240 weeks
  5-year disease progression rate and eGFR slope

OTHER OUTCOMES:
Number of patients with adverse events | Up to 240 weeks
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China